CLINICAL TRIAL: NCT04154501
Title: A Study to Evaluate the Safety and Pharmacokinetics of Single Doses of CNTX-6016 in Healthy Subjects
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of CNTX-6016 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centrexion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CNTX-6016o-HV-101
Record Dates: First submitted 2019-10-07; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Chronic Pain; Nociceptive Pain; Pain
Keywords: Chronic Pain; Nociceptive Pain; Mixed Pain; Cannabinoid; Cannabinoid-2 Receptor Agonist
MeSH Terms: conditions — Chronic Pain; Nociceptive Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- Cohort 1 Placebo (Placebo Comparator): Oral Placebo Capsule
  Interventions: Other: Other: Placebo
- Cohort 1 Drug (Experimental): 25 mg Oral Capsule
  Interventions: Drug: CNTX-6016
- Cohort 2 Placebo (Placebo Comparator): Oral Placebo Capsule
  Interventions: Other: Other: Placebo
- Cohort 2 Drug (Experimental): 50 mg Oral Capsule
  Interventions: Drug: CNTX-6016
- Cohort 3 Placebo (Placebo Comparator): Oral Placebo Capsule
  Interventions: Other: Other: Placebo
- Cohort 3 Drug (Experimental): 100 mg Oral Capsule
  Interventions: Drug: CNTX-6016
- Cohort 4 Placebo (Placebo Comparator): Oral Placebo Capsule
  Interventions: Other: Other: Placebo
- Cohort 4 Drug (Experimental): 300 mg Oral Capsule
  Interventions: Drug: CNTX-6016
- Cohort 5 Placebo (Placebo Comparator): Oral Placebo Capsule
  Interventions: Other: Other: Placebo
- Cohort 5 Drug (Experimental): 450 mg Oral Capsule
  Interventions: Drug: CNTX-6016
- Cohort 6 Placebo (Placebo Comparator): Oral Placebo Capsule
  Interventions: Other: Other: Placebo
- Cohort 6 Drug (Experimental): 600 mg Oral Capsule
  Interventions: Drug: CNTX-6016
- Cohort 7 Placebo (Placebo Comparator): Oral Placebo Capsule
  Interventions: Other: Other: Placebo
- Cohort 7 Drug (Experimental): 800 mg Oral Capsule
  Interventions: Drug: CNTX-6016
- Cohort 9 Placebo (Placebo Comparator): Oral Placebo Capsule
  Interventions: Other: Other: Placebo
- Cohort 9 Drug (Experimental): 1000 mg Oral Capsule
  Interventions: Drug: CNTX-6016
- Cohort 8 Fasted (Experimental): Participant will take 300 mg Oral Capsule in a fasting state, and then fed state.
  Interventions: Drug: CNTX-6016
- Cohort 8 Fed (Experimental): Participant will take 300 mg Oral Capsule in a fed state, and then fasting state.
  Interventions: Drug: CNTX-6016

INTERVENTIONS:
Drug: CNTX-6016 — Oral Dose CNTX-6016
  Arms: Cohort 1 Drug; Cohort 2 Drug; Cohort 3 Drug; Cohort 4 Drug; Cohort 5 Drug; Cohort 6 Drug; Cohort 7 Drug; Cohort 8 Fasted; Cohort 8 Fed; Cohort 9 Drug
Other: Other: Placebo — Oral Dose Placebo
  Arms: Cohort 1 Placebo; Cohort 2 Placebo; Cohort 3 Placebo; Cohort 4 Placebo; Cohort 5 Placebo; Cohort 6 Placebo; Cohort 7 Placebo; Cohort 9 Placebo

SUMMARY:
A Phase 1 double-blind, placebo-controlled, randomized single ascending dose incorporating an open-label, 2-period crossover, food effect cohort.

ELIGIBILITY:
Key Inclusion Criteria:

* Is in good general health as determined by Investigator's review.
* Has a body mass index (BMI) between 18 and 35 kg/m2.
* Non- or ex-smoker (> 1 year) and has not used any nicotine containing products within 12 months prior to screening.
* For females, is not currently pregnant and is either of non-childbearing potential or willing to use an adequate method of birth control.
* For males, must agree to use barrier contraception and not to donate sperm.

Key Exclusion Criteria:

* History of or active cardiac disease, including congestive heart failure, angina, or any arrhythmia.
* Has any history or currently active type of cancer except excised or cured basal cell carcinoma.
* Has a gastrointestinal disorder that could interfere with the absorption of orally administered drugs.
* Has asthma or other severe respiratory disease (e.g., chronic obstructive pulmonary disease) requiring daily prescription medicine.
* Currently has kidney, neurologic, metabolic, or liver disease, or other organ system disease.
* Has a history, current evidence, or is being treated for depression, suicidal ideation, suicide attempt, or any other current psychiatric condition requiring active treatment.
* Has an immunological disorder such as, but not limited to, human immunodeficiency virus (HIV), acquired, or congenital immune deficiency syndrome; autoimmune diseases, such as, but not limited to, rheumatoid arthritis, systemic lupus erythematosus, seronegative spondyloarthropathies or vasculitis, or any infection.
* Has positive screening test for hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Is pregnant, lactating, or planning a pregnancy during the study.
* Has used any prescribed medication within 30 days prior to the first admission or has plans to use any prescribed medication during the study (with the exception of hormonal contraceptives).
* Positive urine screen for alcohol, cotinine, THC and/or drugs of abuse.
* Ingestion of food or beverages containing grapefruit and/or grapefruit juice and/or pomelos during the 7 days prior to dosing and/or during the study period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Safety of single doses of CNTX-6016 - TEAEs | Up to 80 days
  Information regarding treatment emergent adverse events was collected during each dose cohort.
Dose Proportionality of a single doses of CNTX-6016 in healthy subjects | 40 days
  Dose Proportionality of a single doses of CNTX-6016 in healthy subjects.
CNTX-6016 Pharmacokinetics - Cmax | Up to 40 days
  Systemic exposure to CNTX-6016 measured by Cmax.
CNTX-6016 Pharmacokinetics - Tmax | Up to 40 days
  Systemic exposure to CNTX-6016 measured by Tmax.
CNTX-6016 Pharmacokinetics - t1/2 | Up to 40 days
  Systemic exposure to CNTX-6016 measured by t1/2.
CNTX-6016 Pharmacokinetics - AUC 0-t | Up to 40 days
  Systemic exposure to CNTX-6016 measured by AUC 0-t.
CNTX-6016 Pharmacokinetics - AUC 0-inf | Up to 40 days
  Systemic exposure to CNTX-6016 measured by AUC 0-inf.
CNTX-6016 Pharmacokinetics - AUC 0-t/inf | Up to 40 days
  Systemic exposure to CNTX-6016 measured by AUC 0-t/inf.
CNTX-6016 Pharmacokinetics - CL/F | Up to 40 days
  Systemic exposure to CNTX-6016 measured by CL/F.
CNTX-6016 Pharmacokinetics - Vz/F | Up to 40 days
  Systemic exposure to CNTX-6016 measured by Vz/F.
Effect of Gender on CNTX-6016 Pharmacokinetics - Cmax | Up to 80 days
  Effect of Gender on the systemic exposure to CNTX-6016 measured by Cmax.
Effect of Gender on CNTX-6016 Pharmacokinetics - Tmax | Up to 80 days
  Effect of Gender on the systemic exposure to CNTX-6016 measured by tmax.
Effect of Gender on CNTX-6016 Pharmacokinetics - t1/2 | Up to 80 days
  Effect of Gender on the systemic exposure to CNTX-6016 measured by t1/2
Effect of Gender on CNTX-6016 Pharmacokinetics - AUC | Up to 80 days
  Effect of Gender on the systemic exposure to CNTX-6016 measured by AUC.
Effect of Fasted or Fed State on CNTX-6016 Pharmacokinetics - Cmax | Up to 40 days
  Systemic exposure to CNTX-6016 in fasted or fed state as measured by Cmax
Effect of Fasted or Fed State on CNTX-6016 Pharmacokinetics - Tmax | Up to 40 days
  Systemic exposure to CNTX-6016 in fasted or fed state as measured by Tmax
Effect of Fasted or Fed State on CNTX-6016 Pharmacokinetics - t1/2 | Up to 40 days
  Systemic exposure to CNTX-6016 in fasted or fed state as measured by t1/2
Effect of Fasted or Fed State on CNTX-6016 Pharmacokinetics - AUC | Up to 40 days
  Systemic exposure to CNTX-6016 in fasted or fed state as measured by AUC
Urinary Excretion | Up to 6 days
  Urine was collected over a 3-day period (0-72 hrs) in Cohort 8 and analyzed for concentrations of CNTX-6016 in subjects in both the fasted and fed states using Liquid Chromatography Mass Spectrometry.

SECONDARY OUTCOMES:
Plasma and Urine Metabolite Mining | 5 days
  Urine was collected over a 3-day period (0-72hrs) in Cohort 9 (1000mg) and analyzed for concentrations of parent and metabolites of CNTX-6016 using Liquid Chromatography Mass Spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Randall M Stevens, MD, Study Chair — Centrexion Therapeutics
Locations (1):
- Altasciences Clinical Research, Overland Park, Kansas, United States